CLINICAL TRIAL: NCT01450137
Title: A Phase II, Randomized, Double-blind, Placebo Controlled Study of Tocilizumab in Patients With Giant Cell Arteritis
Brief Title: Tocilizumab for Patients With Giant Cell Arteritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: University of Bern (Other); Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 168/10
Record Dates: First submitted 2011-10-03; First posted 2011-10-12 (Estimated); Results first posted 2019-02-12 (Actual); Last update posted 2019-02-12 (Actual); Status verified 2018-09

CONDITIONS: Giant Cell Arteritis
Keywords: Giant Cell Arteritis; Tocilizumab; Antibodies, Monoclonal; Glucocorticoids
MeSH Terms: conditions — Giant Cell Arteritis | interventions — tocilizumab; Glucocorticoids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tocilizumab (Experimental): Tocilizumab 8mg/kg every 4 weeks until week 52.
  Interventions: Drug: Tocilizumab + Glucocorticoids (GCs)
- Placebo (Placebo Comparator): Placebo every 4 weeks until week 52.
  Interventions: Drug: Placebo + Glucocorticoids (GCs)

INTERVENTIONS:
Drug: Tocilizumab + Glucocorticoids (GCs) — Tocilizumab 8mg/kg every 4 weeks until week 52.
  Arms: Tocilizumab
Drug: Placebo + Glucocorticoids (GCs) — Placebo every 4 weeks until week 52.
  Arms: Placebo

SUMMARY:
Giant-cell arteritis (GCA) is an immune-mediated disease that mostly affects people older than 50 years of age. Glucocorticoid (GC) treatment dramatically alters the symptoms and course of GCA, reducing the likelihood of vascular complications that could lead e.g. to blindness. However, relapses usually occur when GC dosages are tapered, resulting in frequent re-treatment with high cumulative dosages of GC over time with substantial toxicity and morbidity (e.g. diabetes mellitus, infections, enhanced cardiovascular risk, osteoporotic fractures, cataracts).

Therefore, novel therapies are needed that effectively reduce the dose and duration of GC treatment and provide more durable remissions of GCA.

Tocilizumab (TCZ) is a humanized monoclonal antibody directed against the human interleukin-6 receptor (IL-6R). Elevated tissue and serum levels of IL-6 have been implicated in giant cell arteritis. Inhibition of IL-6 and/or its receptor therefore represents a new and novel approach for the treatment of RA.

The primary endpoint is the proportion of patients that have achieved complete remission of disease after treatment with TCZ compared to treatment with placebo at week 12. All patients will receive glucocorticoids in a standardized form.

DETAILED DESCRIPTION:
Background

Giant-cell arteritis (GCA) is an immune-mediated disease that mostly affects people older than 50 years of age. Glucocorticoid (GC) treatment dramatically alters the symptoms and course of GCA, reducing the likelihood of vascular complications that could lead e.g. to blindness. However, relapses usually occur when GC dosages are tapered, resulting in frequent re-treatment with high cumulative dosages of GC over time with substantial toxicity and morbidity (e.g. diabetes mellitus, infections, enhanced cardiovascular risk, osteoporotic fractures, cataracts).

Therefore, novel therapies are needed that effectively reduce the dose and duration of GC treatment and provide more durable remissions of GCA.

Tocilizumab (TCZ) is a humanized monoclonal antibody directed against the human interleukin-6 receptor (IL-6R). Elevated tissue and serum levels of IL-6 have been implicated in giant cell arteritis. Inhibition of IL-6 and/or its receptor therefore represents a new and novel approach for the treatment of RA.

Objective

The primary endpoint is the proportion of patients that have achieved complete remission of disease (normal ESR and CRP + absence of signs and symptoms) at Week 12 at a GC dose of 0.1 mg/kg/d of prednisone.

Methods

2-arm (Tocilizumab + Glucocorticoids (GCs) vs. Placebo + GCs), randomized, placebo-controlled, double blind, monocentric trial in patients with newly onset or relapsing giant cell arteritis (GCA), satisfying ACR criteria AND an elevated sedimentation rate above 40 mm/h and a CRP > 20 mg/L AND a biopsy proven GCA OR a large vessel vasculitis assessed by MR Angiography (MRA).

ELIGIBILITY:
Inclusion Criteria:

* Patients with newly onset or relapsed GCA
* > 50 years of age
* satisfying ACR criteria
* elevated sedimentation rate above 40 mm
* CRP > 20 mg/L
* Patients with histologically proven GCA or with large vessel vasculitis assessed by MRI

Exclusion Criteria

* Rheumatic diseases (except for CPPD/chondrocalcinosis) other than GCA/Takayasu disease or polymyalgia rheumatica (i.e., RA, autoimmune connectivitides, other systemic vasculitides, a.o.)
* Evidence of significant and/or uncontrolled concomitant disease
* Diagnosis of GCA > 4 weeks before screening visit and beginning of GC treatment > 4 weeks before screening (only valid for new onset GCA), or when a patient received treatment with tocilizumab or with other biological agents (such as TNFα-blockers) within 3 months before screening
* Any condition or general state of health which, in the Investigator's opinion, would preclude participation in the study
* Actual or recent myocardial infarction (within the last 3 months before screening visit)
* Significant cardiac disease (NYHA Class III and IV), known severe chronic obstructive pulmonary disease (COPD) (FEV1 < 50% predicted or Functional dyspnoea > Grade 3 on the MRC Dyspnoea Scale) or other significant pulmonary disease
* Uncontrolled disease (such as asthma, psoriasis or inflammatory bowel disease) where flares are commonly treated with oral or injectable corticosteroids
* Known active infection of any kind, or any major episode of infection requiring hospitalization or treatment with i.v. anti-infectives within 4 weeks of baseline or completion of oral anti-infectives within 2 weeks prior to baseline
* History of deep space/tissue infection (e.g. fasciitis, abscess, osteomyelitis) within 52 weeks prior to baseline
* Any surgical procedure, including bone/joint surgery within 8 weeks prior to baseline or planned within the duration of the study
* History of serious recurrent or chronic infection (for screening for a chest infection a chest radiograph will be performed at screening if not performed within 12 weeks prior to screening)
* Lack of peripheral venous access
* Body weight > 150 kg or BMI > 35
* Previous treatment with tocilizumab or any other biological agent
* Treatment with any investigational agent within 28 days of screening or 5 half-lives of the investigational drug (whichever is the longer)
* History of severe allergic or anaphylactic reaction to any biologic agent or known hypersensitivity to any component of tocilizumab (RoActemra)
* Receipt of any vaccine within 28 days prior to baseline (a patient's vaccination record and need for immunization prior to receiving tocilizumab/placebo must be carefully investigated)
* Positive tests for hepatitis B surface antigen (HBsAg), Hepatitis B core antibody (HbcAb) or hepatitis C serology
* Positive Quantiferon-TB® test for latent Tb without subsequent INH prophylaxis
* Patients with active Tb which had to be treated for Tb within 2 years before the screening visit

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2011-09; Primary Completion 2014-12 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Villiger, Prof, Principal Investigator — Department of Rheumatology, Clinical Immunology Allergology, University Hospital, Inselspital; Michael Seitz, Prof, Principal Investigator — Department of Rheumatology, Clinical Immunology Allergology, University Hospital, Inselspital
Locations (1):
- Department of Rheumatology, Clinical Immunology Allergology, University Hospital, Inselspital, Bern, Switzerland

REFERENCES:
- [Result] Villiger PM, Adler S, Kuchen S, Wermelinger F, Dan D, Fiege V, Butikofer L, Seitz M, Reichenbach S. Tocilizumab for induction and maintenance of remission in giant cell arteritis: a phase 2, randomised, double-blind, placebo-controlled trial. Lancet. 2016 May 7;387(10031):1921-7. doi: 10.1016/S0140-6736(16)00560-2. Epub 2016 Mar 4. PMID 26952547
- [Derived] Gloor AD, Yerly D, Adler S, Reichenbach S, Kuchen S, Seitz M, Villiger PM. Immuno-monitoring reveals an extended subclinical disease activity in tocilizumab-treated giant cell arteritis. Rheumatology (Oxford). 2018 Oct 1;57(10):1795-1801. doi: 10.1093/rheumatology/key158. PMID 29961816

RESULTS

PARTICIPANT FLOW:
Period: Up to Week 12
Arm/Group | Tocilizumab | Placebo
Started | 20 | 10
Completed | 18 | 7
Not Completed | 2 | 3
Not completed — Adverse Event | 2 | 1
Not completed — Withdrawal by Subject | 0 | 2
Period: Week 12 to Study End
Arm/Group | Tocilizumab | Placebo
Started | 18 | 7
Completed | 18 | 5
Not Completed | 0 | 2
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tocilizumab | Placebo | Total
Number analyzed (Participants) | 20 | 10 | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.3 (8.9) | 68.8 (16.9) | 70.5 (11.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 8 | 21
  Male | 7 | 2 | 9
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (3.0) | 27.9 (3.7) | 25.0 (3.8)
New onset giant cell arteritis [Count of Participants; unit: Participants] | 16 | 7 | 23
Biopsy of the temporal artery [Count of Participants; unit: Participants]
  Normal | 5 | 0 | 5
  Abnormal | 13 | 8 | 21
  Not done | 2 | 2 | 4
Thoracoabdominal MR angiography [Count of Participants; unit: Participants]
  Normal | 9 | 2 | 11
  Abnormal | 11 | 6 | 17
  Not done | 0 | 2 | 2
Symptoms and signs of giant cell arteritis [Count of Participants; unit: Participants]
  Fever >= 38°C | 1 | 1 | 2
  Weight loss > 2kg within 4 weeks | 6 | 3 | 9
  Night sweats | 3 | 2 | 5
  Headache | 13 | 5 | 18
  Scalp tenderness | 9 | 1 | 10
  Claudication of tongue | 2 | 0 | 2
  Masseter muscle claudication | 11 | 4 | 15
  Claudication of upper limbs | 4 | 2 | 6
  Claudication of lower limbs | 0 | 2 | 2
  Visual impairment | 5 | 2 | 7
Blood pressure [Mean (Standard Deviation); unit: mmHg] — Population: Missing data.
  mmHg
    Systolic right arm: number analyzed (Participants) | 20 | 9 | 29
    Systolic right arm | 130.6 (18.0) | 137.7 (16.4) | 132.8 (17.5)
    Diastolic right arm: number analyzed (Participants) | 20 | 9 | 29
    Diastolic right arm | 74.3 (11.8) | 77.7 (15.2) | 75.3 (12.8)
    Systolic left arm: number analyzed (Participants) | 19 | 8 | 27
    Systolic left arm | 131.3 (16.3) | 136.9 (13.0) | 132.9 (15.3)
    Diastolic left arm: number analyzed (Participants) | 19 | 8 | 27
    Diastolic left arm | 75.1 (11.5) | 82.8 (8.5) | 77.3 (11.1)
Erythrocyte sedimentation rate [Median (Inter-Quartile Range); unit: mm/h] | 69.0 [45.5 to 80.0] | 40.0 [27.3 to 68.8] | 54.5 [40.0 to 80.0]
C-reactive protein [Median (Inter-Quartile Range); unit: mg/L] | 25.5 [16.8 to 50.3] | 39.0 [23.5 to 64.3] | 31.5 [19.8 to 54.3]

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients That Have Achieved Complete Remission of Disease
Time Frame: 12 weeks
Population: All randomized patients, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 20 | 10
Participants | 17 | 4
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.0301, Fisher Exact; Risk Difference (RD) = 0.45, 95% CI 2-sided [0.11 to 0.79]

2. Secondary Outcome: Number of Relapse Free Patients
Time Frame: 12 months
Population: All randomized patients, intention-to-treat
Measure: Count of Participants; unit: Participants
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 20 | 10
Participants | 17 | 2
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.0010, Fisher Exact; Risk Difference (RD) = 0.65, 95% CI 2-sided [0.36 to 0.94]

3. Secondary Outcome: Cumulative Dose of GCs in mg/kg
Description: cumulative weight-adapted prednisolone dose
Time Frame: 12 months
Population: All randomized patients, intention-to-treat
Measure: Median (Inter-Quartile Range); unit: mg/kg
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 20 | 10
mg/kg | 43 [39 to 52] | 110 [88 to 150]
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.0005, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Restricted Mean Survival Time to First Relapse After Induction of Remission
Time Frame: 12 months
Population: All randomized patients, intention-to-treat
Measure: Mean (95% Confidence Interval); unit: Weeks
Arm/Group | Tocilizumab | Placebo
Number analyzed (Participants) | 20 | 10
Weeks | 50 [46 to 54] | 25 [11 to 38]
Statistical Analysis 1: Comparison: Tocilizumab vs Placebo; Test type: Superiority; p = 0.0005, z-test; Mean Difference (Final Values) = 25, 95% CI 2-sided [11 to 39] — Difference between restricted mean survival time at 12 months

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tocilizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 1/10
Serious Adverse Events (participants affected / at risk) | 7/20 | 5/10
Other Adverse Events (participants affected / at risk) | 11/20 | 6/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=20) | Placebo (N=10)
Gastrointestinal disease (Gastrointestinal disorders) | 3 (3) | 1 (1)
Cardiovascular disease (Cardiac disorders) | 1 (1) | 2 (3)
Osteoporotic fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
Glucocorticoid related hyperglycaemia and myopathia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Infectious disease (Infections and infestations) | 1 (1) | 0 (0)
Skin disease (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tocilizumab (N=20) | Placebo (N=10)
Cardiovascular disease (Cardiac disorders) | 0 (0) | 2 (2)
Cystic lesion mamma (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Gastrointestinal disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Glucocorticoid-related hyperglycaemia and myopathia (Blood and lymphatic system disorders) | 1 (2) | 1 (1)
Infectious disease (Infections and infestations) | 7 (9) | 1 (1)
Musculoskeletal disease (Musculoskeletal and connective tissue disorders) | 4 (5) | 3 (6)
Osteoporotic fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Skin disease (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes